CLINICAL TRIAL: NCT03413865
Title: A Pilot Study of a Nurse and Pharmacist Led OTN (Ontario Telemedicine Network) Based Clinic for Management of Prostate Cancer Patients on Oral Therapy
Brief Title: Telemedicine Clinic for Prostate Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grand River Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OTN Study
Record Dates: First submitted 2018-01-12; First posted 2018-01-29 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Cancer, Treatment-Related
MeSH Terms: conditions — Neoplasms, Second Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OTN virtual clinic (Experimental): Pharmacist and nurse led OTN based remote teleconference based clinic (OTN) The OTN clinic will be conducted by providing the patient with a link via email which will allow the patient to access OTN teleconferencing and meet virtually with a pharmacist and nurse during a previously scheduled appointment. Virtual clinic appointments will be 30 minutes long and will consist of a patient assessment and open ended questions about the patient health status using a modified version of the validated MOATT (MASCC Oral Agent Teaching Tool) created by the Multidisciplinary Association of Supportive Care in Cancer.
  Interventions: Other: Visits conducted via Telemedicine
- In person Visits (No Intervention): Patients are followed in person at the cancer clinic based on standard of care guidelines

INTERVENTIONS:
Other: Visits conducted via Telemedicine — Patients will be followed via telemedicine with visits lead by a Pharmacist and a Nurse
  Arms: OTN virtual clinic

SUMMARY:
This randomized, open label study will evaluate a nurse and pharmacist led clinic conducted remotely from Grand River Regional Cancer Centre at Grand River Hospital (GRRCC/GRH) using OTN teleconferencing as a platform for patients with prostate cancer receiving oral chemotherapy agents.

ELIGIBILITY:
Inclusion Criteria:

1. Male over 18 years of age with prostate cancer receiving oral treatment with abiraterone or enzalutamide.
2. Ability to provide consent to study.
3. Willingness to complete study questionnaires and a semi-structured exit interview.
4. Adequate command of the English language to complete study questionnaire and survey.
5. Access to technology to allow a link to the virtual telemedicine clinic. (excluding control group)
6. Willingness to participate in videoconference with pharmacist or nurse from their home environment. (excluding control group)

Exclusion Criteria:

1. Patients receiving oral anti-cancer therapy other than abiraterone and enzalutamide.
2. Patients lacking the technology at home to participate in the virtual telemedicine clinic. (excluding control group)

   -

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate Cancer Patients
Enrollment: 80 (Estimated)
Dates: Start 2016-10-28 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction with overall care | 2 Years
  The primary outcome will be a comparison of patient satisfaction with overall care utilizing a validated scale between the group of patients using the OTN clinic and a group of control patients receiving conventional care at GRRCC

CONTACTS AND LOCATIONS:
Locations (1):
- Grand River Hospital, Kitchener, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No